CLINICAL TRIAL: NCT03664596
Title: Evaluation Of The Therapeutic And Dietary Properties Of The Sublimated Mare's Milk Supplement In Patients With Non-Alcoholic Steatohepatitis
Brief Title: Therapeutic And Dietary Effects Of The Sublimated Mare's Milk Supplement In Patients With Non-Alcoholic Steatohepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Centre Hospital of the President's Affairs Administration, Republic of Kazakhstan (Other Government)
Collaborators: Eurasia Invest Ltd. (Industry); Ministry of Education and Science, Republic of Kazakhstan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDP.NAS.01
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: Non-alcoholic Steatohepatitis; Mare milk; Immune markers
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary supplement only (Experimental): Participants will take a sublimated mare milk of 1 sachet 3 times a day during 2 months.
  Interventions: Dietary Supplement: Sublimated mare's milk
- Dietary supplement and ursodeoxycholic acid therapy (Other): Patients with non-alcoholic steatohepatitis will take ursodeoxycholic acid (2-3 times/day) combined with the mare's milk supplement (1 sachet, 3 times/day) for two months.
  Interventions: Dietary Supplement: Sublimated mare's milk; Drug: Ursodeoxycholic Acid
- Ursodeoxycholic acid therapy only (Active Comparator): Patients with verified diagnosis of non-alcoholic steatohepatitis would be given treatment of ursodeoxycholic acid (2-3 times/day) for a two-month period.
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Dietary Supplement: Sublimated mare's milk — Supplement obtained through sublimation of mare milk, packed into one-dosage sachet (20g), and dissolved in a warm water (36 degrees of Celcius).
  Arms: Dietary supplement and ursodeoxycholic acid therapy; Dietary supplement only
Drug: Ursodeoxycholic Acid — Ursodeoxycholic acid in the form of 250 mg capsule.
  Arms: Dietary supplement and ursodeoxycholic acid therapy; Ursodeoxycholic acid therapy only

SUMMARY:
This study evaluates the dietary and therapeutic effect of supplement consisting of sublimated mare milk among patients with non-alcoholic steatohepatitis.

DETAILED DESCRIPTION:
Nonalcoholic steatohepatitis (NASH) is characterized by the liver damage in the form of fatty degeneration and hepatitis in people who do not abuse alcohol. The disease often develops in middle-aged women with excessive body weight, increased blood glucose and blood lipids, but can occur in all age groups and in both sexes. In most cases, the disease is asymptomatic. Laboratory data indicate an increase in the level of aminotransaminases. Ultrasound reveals hyperechoic tissue of the liver due to diffuse fatty infiltration. The degree of steatosis can also be estimated by a controlled attenuation parameter (CAP - Controlled Attenuation Parameter) in the fibroelastometry of liver tissue. It is also possible to verify the degree of fibrosis of liver tissue in its presence. Given that the mare's milk has therapeutic and dietary properties for various diseases of the internal organs, including liver diseases, the investigators decided to study its therapeutic effectiveness in NASH.

In this clinical study, the effectiveness of mare's milk in NASH will be studied in comparison with control groups taking monotherapy with ursodeoxycholic acid (UDCA) and combined therapy (mare's milk and UDCA). Patients will receive a sublimated form of mare's milk in the appropriate dosage within 2 months, and the results of clinical laboratory and instrumental studies will be compared among themselves using statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a verified diagnosis of non-alcoholic steatohepatitis;
* Aged 16 to 60 years;
* Absence of an allergic reaction to dairy products;
* Willingness to consent to participate in the study.
* Consent to adhere to treatment

Exclusion Criteria:

* Taking antibiotics, cytostatics and steroids during the last 3 months;
* Taking alcohol hepatotoxic doses (no more than 30 g alcohol per day for men and not more than 20 g for women);
* History of oncological diseases;
* Presence of diabetes mellitus, decompensated forms of diseases, intestinal dyspepsia, hypertension (blood pressure 140/90 mm Hg and more at the time of the initial visit to the doctor), tuberculosis;
* A positive result of screening for antibodies to viral hepatitis B, C and D, as well as HIV
* Presence of concomitant diseases of the kidneys, liver, cardiovascular, respiratory and other body systems, oncological, mental health and decompensated endocrine diseases, tuberculosis, and HIV infection;
* Pregnancy and/or lactation;
* Patient involvement in other clinical trials within the last 3 months;
* Refusal to participate in the study.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in liver function indicators | Baseline, Week 2, Week 4, Week 6, Week 8
  Blood samples will be taken to determine changes in bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase AST, gamma-glutamyl transpeptidase (GGTP), alkaline phosphatase,
Change in degree of steatosis and fibrosis (fibroelastometry method). | Baseline, Week 8
  Degree of steatosis and fibrosis will evaluated via fibroelastometry method.
Change in degree of steatosis and fibrosis (ultrasound method) | Baseline, Week 8
  Ultrasound will be used for assessment of steatosis and fibrosis.

SECONDARY OUTCOMES:
Change in biochemical blood test results (cholesterol, glucose) | Baseline, Week 2, Week 4, Week 6, Week 8
  Proportion of those with deviations from normal range will be reported and compared across periods and groups.
Change in weight. | Baseline, Week 2, Week 4, Week 6, Week 8
  Frequency of patients with decreased weight will be detected and compared across groups/periods.
Detection of general clinical symptoms of non-alcoholic steatohepatitis. | Baseline, Week 2, Week 4, Week 6, Week 8
  Symptoms such as of malaise, abdominal discomfort, vague right upper quadrant abdominal pain will be identified in patients during physical examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Centre Hospital of the President's Affairs Administration, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sidhu GS, Brown MA, Johnson AR. Autoxidation in milk rich in linoleic acid. I. An objective method of measuring autoxidation and evaluating antioxidants. J Dairy Res. 1975 Feb;42(1):185-95. doi: 10.1017/s0022029900015211. PMID 1123470
- [Background] Sidhu GS, Brown MA, Johnson AR. Autoxidation in milk rich in linoleic acid. II. Modification of the initiation system and control of oxidation. J Dairy Res. 1976 Jun;43(2):239-50. doi: 10.1017/s002202990001579x. PMID 956472
- [Background] Rong J, Zheng H, Liu M, Hu X, Wang T, Zhang X, Jin F, Wang L. Probiotic and anti-inflammatory attributes of an isolate Lactobacillus helveticus NS8 from Mongolian fermented koumiss. BMC Microbiol. 2015 Oct 2;15:196. doi: 10.1186/s12866-015-0525-2. PMID 26428623
- [Background] Aryantini NP, Yamasaki E, Kurazono H, Sujaya IN, Urashima T, Fukuda K. In vitro safety assessments and antimicrobial activities of Lactobacillus rhamnosus strains isolated from a fermented mare's milk. Anim Sci J. 2017 Mar;88(3):517-525. doi: 10.1111/asj.12668. Epub 2016 Aug 1. PMID 27476815
- [Background] Ma YY, Li L, Yu CH, Shen Z, Chen LH, Li YM. Effects of probiotics on nonalcoholic fatty liver disease: a meta-analysis. World J Gastroenterol. 2013 Oct 28;19(40):6911-8. doi: 10.3748/wjg.v19.i40.6911. PMID 24187469
- [Background] Zhang B, Lu XL, Song YH, Shi HT, Li J, Geng Y. [Changes in the intestinal microenvironment during development of alcoholic fatty liver disease and related effects of probiotic therapy]. Zhonghua Gan Zang Bing Za Zhi. 2012 Nov;20(11):848-52. doi: 10.3760/cma.j.issn.1007-3418.2012.11.010. Chinese. PMID 23206305
- [Background] Valiev AG, Valieva TA, Valeeva GR, Speranskii VV, Levachev MM. [The effect of the essential fatty acids in mare's milk on the function of the immune system and of nonspecific resistance in rats]. Vopr Pitan. 1999;68(3):3-6. Russian. PMID 10392421
- [Background] Abdel-Salam AM, Al-Dekheil A, Babkr A, Farahna M, Mousa HM. High fiber probiotic fermented mare's milk reduces the toxic effects of mercury in rats. N Am J Med Sci. 2010 Dec;2(12):569-75. doi: 10.4297/najms.2010.2569. PMID 22558569
- [Background] Guri A, Paligot M, Crevecoeur S, Piedboeuf B, Claes J, Daube G, Corredig M, Griffiths MW, Delcenserie V. In vitro screening of mare's milk antimicrobial effect and antiproliverative activity. FEMS Microbiol Lett. 2016 Jan;363(2):fnv234. doi: 10.1093/femsle/fnv234. Epub 2015 Dec 9. PMID 26656278
- [Result] Oshakbayev K, Bimbetov B, Manekenova K, Bedelbayeva G, Mustafin K, Dukenbayeva B. Severe nonalcoholic steatohepatitis and type 2 diabetes: liver histology after weight loss therapy in a randomized clinical trial. Curr Med Res Opin. 2019 Jan;35(1):157-165. doi: 10.1080/03007995.2018.1547696. Epub 2018 Nov 28. PMID 30431378
- [Result] Bimbetov B., Zhangabylov A., Aitbaeva S., Rakhimzhanova M, Bakytzhanuly A. The result of taking mare's milk for nonalcoholic steatohepatitis // Journal of Global Pharma Technology. Volume 11 Issue 08 (2019) August 2019. -Р.268-273.
- [Result] Bimbetov B., Zhangabylov A., Aitbaeva S., Bakytzhanuly A., Utepbergenova G. Use of the mare's milk of the treatment of non-alcoholic steatohepatitis // Systematic Reviews in Pharmacy. -2020.